CLINICAL TRIAL: NCT04897113
Title: Multicenter, Open, Prospective, Randomized Trial of Efficacy and Safety of the Plasmapheresis Method With Albumin Compensation Compared With the Plasmapheresis Method Without Albumin Compensation for Aging Biomarkers Correction in Men and Women Aged 40 to 55 Years Old
Brief Title: Study of Efficacy and Safety of the Plasmapheresis Method With Albumin Compensation Compared With the Plasmapheresis Method Without Albumin Compensation for Aging Biomarkers Correction in Men and Women Aged 40 to 55 Years Old
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Medical Research Center for Rehabilitation and Balneology (Other)
Collaborators: The Orenburg Regional Clinical Hospital (Other Government); DNKOM LLC (Other); Pirogov Russian National Research Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RU-RB-01-01-21 of 08.02.2021
Record Dates: First submitted 2021-05-18; First posted 2021-05-21 (Actual); Last update posted 2021-05-21 (Actual); Status verified 2021-05

CONDITIONS: Hypercholesterolemia; Hyperbilirubinemia; Hyper IgE Syndrome; Hyper Beta Lipoproteinemia; Hyper Eosinophilic Syndrome; Hyper-LDL-cholesterolemia; Gout; Diabetes; Nervous System Diseases; Neuromuscular Diseases; Cardiovascular Diseases; Urologic Diseases
Keywords: plasmapheresis; plasma exchange; albumin; biomarkers of aging; age-related diseases
MeSH Terms: conditions — Hypercholesterolemia; Hyperbilirubinemia; Job Syndrome; Hyperlipoproteinemia Type II; Hypereosinophilic Syndrome; Gout; Diabetes Mellitus; Nervous System Diseases; Neuromuscular Diseases; Cardiovascular Diseases; Urologic Diseases | interventions — Plasma Exchange; Albumins; Plasmapheresis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- plasmapheresis with albumin compensation (Experimental): a course of hardware plasmapheresis procedures with replacement by colloidal (5% albumin solution) and crystalloid solutions (saline) in a ratio of 1: 3
  Interventions: Procedure: plasma exchange with albumin
- plasmapheresis without albumin compensation (Experimental): a course of hardware plasmapheresis procedures without replacement by albumin solution, only crystalloid solutions (saline).
  Interventions: Procedure: plasma exchange without albumin

INTERVENTIONS:
Procedure: plasma exchange with albumin — plasma exchange with albumin, two per week, 110% of the circulating plasma volume
  Other Names: plasmapheresis with albumin
  Arms: plasmapheresis with albumin compensation
Procedure: plasma exchange without albumin — plasma exchange without albumin, two per week, 110% of the circulating plasma volume
  Other Names: plasmapheresis without albumin
  Arms: plasmapheresis without albumin compensation

SUMMARY:
Reaching active aging makes it important to implement new methods affecting the biological age of a person. Biochemical parameters of a blood test are aging biomarkers that are ones of the most accessible for testing. We know that, with age, there is increase in levels of LDL, triglycerides, homocysteine and other biomarkers relating the body state.

Methods of extracorporeal hemocorrection showed good results in this area. For instance, the use of plasmapheresis is very effective during prophylaxis, treatment and rehabilitation after various diseases/injuries. The main effects of plasmapheresis are related to removal of endo- and exotoxins, including products of lipid peroxidation, and to draining effect as a result of a heavy flow of interstitial fluid containing products of pathometabolism into the blood stream within concentration gradient (by "dynamic equilibrium" in concentration of different substances in intracellular, interstitial and intravascular compartments). These effects are also related to release of receptors, their sensitization to their own neurohumoral regulation mechanisms, to insulin, in particular (as consequences, lower glucose tolerance, lower substrate glycation).

DETAILED DESCRIPTION:
Reaching active aging makes it important to implement new methods affecting the biological age of a person. Biochemical parameters of a blood test are aging biomarkers that are ones of the most accessible for testing. We know that, with age, there is increase in levels of LDL, triglycerides, homocysteine and other biomarkers relating the body state.

One of the initial approaches of anti-ageing therapy is detoxification, reocorrection and immunocorrection. Methods of extracorporeal hemocorrection showed good results in this area. For instance, the use of plasmapheresis is very effective during prophylaxis, treatment and rehabilitation after various diseases/injuries. The main effects of plasmapheresis are related to removal of endo- and exotoxins, including products of lipid peroxidation, and to draining effect as a result of a heavy flow of interstitial fluid containing products of pathometabolism into the blood stream within concentration gradient (by "dynamic equilibrium" in concentration of different substances in intracellular, interstitial and intravascular compartments). These effects are also related to release of receptors, their sensitization to their own neurohumoral regulation mechanisms, to insulin, in particular (as consequences, lower glucose tolerance, lower substrate glycation).

Thus, at this stage, experts assess effectiveness and organize data of existing prevention methods for premature aging and correction of aging biomarkers, as well as develop comprehensive programs for drug-free and pharmacological intervention. Introduction of the body detoxification method based on extracorporeal hemocorrection (developed in FGBU Russian Scientific Center for Medical Rehabilitation and Balneology of Ministry of Health of Russian Federation) may extend the range of effective and safe methods within such programs, as well as lower patients' biological age and, thus, lower risks of developing age-related diseases, decrease number of disability cases, which can contribute to life prolonging and improvement of its quality.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Men and women aged 40-55.
* Body mass index <30 kg / m2.
* Level increase of one or several aging markers.
* Understanding of requirements for study participants, written consent to participate in the study (including volunteer's consent for his/her health information related to the study to be used and passed on) and to perform procedures outlined in study protocol.
* Negative pregnancy test for women of childbearing potential.

Non-inclusion Criteria:

* Refusal to participate in the study.
* Any health conditions that, according to investigators, might prevent volunteers from participating in the study.
* Mental disorders, past medical history included.
* 10 + alcohol units per week (one alcohol unit equals 0,5 l of beer, 200 ml of wine or 50 ml of hard liquors) or any records of alcohol addiction.
* Drug addiction, chemical abuse.
* Pregnancy or breastfeeding.
* Past medical history of severe allergic reactions.
* General contraindications to plasmapheresis procedures.
* Any other health conditions or reasons that, according to investigators, might increase risks for participants or reduce the likelihood of results needed to meet the study goals.

Exclusion Criteria:

* Voluntary refusal to participate in the study.
* Investigator doctor's decision on participant's exclusion for this participant's own benefit.
* Participant refuses to cooperate with investigator or is undisciplined.
* In case participant misses one or several study procedures or follow-up visits.
* Development of severe adverse reactions or severe diseases/conditions unrelated to the study, requiring withdrawal from therapy.
* Positive pregnancy test.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-05-12 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Dynamics summary for improvement of aging biomarkers' values assessed by a patient's biochemical blood count | 1 month
  Dynamics summary for improvement of aging biomarkers' values assessed by a patient's biochemical blood count at visit 6, compared with initial values (visit 0).

SECONDARY OUTCOMES:
Dynamics summary for improvement of aging biomarkers' values assessed by a patient's biochemical blood count | 17 (+/- 2) days
  Dynamics summary for aging biomarkers' values assessed by a patient's biochemical blood count at visit 5, compared with initial values (visit 0).
Dynamics summary for aging biomarkers' values assessed by a patient's complete blood count | 1 month
  Dynamics summary for aging biomarkers' values assessed by a patient's complete blood count at visits 5 and 6, compared with initial values (visit 0).
Dynamics summary for aging biomarkers' values assessed by a patient's blood serological test | 1 month
  Dynamics summary for aging biomarkers' values assessed by a patient's blood serological test at visits 5 and 6, compared with initial values (visit 0).
Dynamics summary for aging biomarkers' values assessed by a patient's coagulation test | 1 month
  Dynamics summary for aging biomarkers' values assessed by a patient's coagulation test at visits 5 and 6, compared with initial values (visit 0).
Dynamics of results according to the method of "phenotypic age" | 1 month
  Dynamics of results according to the method of "phenotypic age" assessment with the use of values of complete and biochemical blood counts at visits 5 and 6, compared with initial values (visit 0).
  An assessment of the "phenotypic age" will be carried out (Morgan E. et al., 2018). For counting, 10 markers are used: albumin, creatinine, glucose, C-reactive protein, percentage of lymphocytes, average cell volume, distribution width of erythrocytes, alkaline phosphatase, leukocyte count, chronological age.
Dynamics of results according to the method of biological age | 1 month
  Dynamics of results according to the method of biological age assessment with the use of values of complete and biochemical blood counts at visits 5 and 6, compared with initial values (visit 0). The biological age will be assessed by the method of Putin E., Mamoshina P. et al., 2016. The following markers are used for calculation by this method: albumin, glucose, urea, cholesterol, total protein, sodium, creatinine, hemoglobin, total bilirubin, triglycerides , HDL cholesterol, LDL cholesterol (Friedewald), calcium, potassium, hematocrit, MCHC, MCV, platelets, erythrocytes (erythrocytes), weight, height.
  An online system available at http://www.aging.ai will be used to estimate biological age.
Dynamic pattern according to ECG results | 1 month
  Dynamic pattern according to ECG results in 12 leads at visits 5 and 6, compared with initial values (visit 0).
Dynamic pattern according to results of vascular ultrasonography | 1 month
  Dynamic pattern according to results of vascular ultrasonography at visits 5 and 6, compared with initial values (visit 0).
SF-36 scale | 1 month
  Change of scores according to every scale out of all 8 scales from the SF-36 questionnaire at visits 5, 6 and 7, compared with initial values (visit 0).
HAM questionnaire | 1 month
  Dynamics of subjective assessment of a patient's current psycho emotional state (HAM questionnaire) at visits 5, 6 and 7, compared with initial values (visit 0). The Hamilton Rating Scale for Depression (HRSD), also called the Hamilton Depression Rating Scale (HDRS), abbreviated HAM-D, is a multiple-item questionnaire used to provide an indication of depression, and as a guide to evaluate recovery.
scales of the "Health-Promoting Lifestyle Profile" | 1 month
  Change of scores according to every scale out of 6 scales of the "Health-Promoting Lifestyle Profile" questionnaire at visits 5, 6 and 7, compared with initial values (visit 0).

CONTACTS AND LOCATIONS:
Overall Officials: Ilmira Gilmutdinova, Study Chair — Federal State Budgetary Institution "National Medical Center for Rehabilitation and Balneology" of the Ministry of Health of Russia
Locations (2):
- Russia (2):
  - Federal State Budgetary Institution "National Medical Center for Rehabilitation and Balneology" of the Ministry of Health of Russia, Moscow
  - Orenburg regional clinical blood transfusion station, Orenburg